CLINICAL TRIAL: NCT00256165
Title: Left Ventricular Regression European Study
Brief Title: REST Study: Left Ventricular Regression European Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Christophe Bailleul, St. Jude Medical
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CS04009TV
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Tissue valve — Aortic valve replacement

SUMMARY:
The purpose of this study is to obtain data regarding the left ventricular mass (LVM) regression 6 months after the implant of an SJM Epic™ and SJM Epic™ Supra valve by comparing LVM regression measured with magnetic resonance imaging (MRI) to LVM regression measured with echocardiography (2-dimensional [2D] mandatory; 3-dimensional [3D] in sites where the technology is available).

ELIGIBILITY:
Inclusion Criteria:

* Patient requires, for the first time, isolated aortic valve replacement due to aortic stenosis or mixed aortic stenosis disease etiology when aortic stenosis is predominant and aortic regurgitation is mild.
* Patient is of legal age in the host country.
* Patient (or legal guardian) has signed a study specific informed consent form

Exclusion Criteria:

* Patient was previously operated on with any heart surgery including heart valve replacement or coronary artery bypass graft (CABG); or underwent any form of myocardial revascularization in the past (including stents), etc.
* Patient requires any concomitant heart surgery other than the isolated native aortic heart valve replacement and concomitant ascending aortic replacement (e.g not allowed are: multiple valve replacements or concomitant CABG, pacemaker insertions, or severe septal hypertrophy needing surgical excision, etc.)
* Patient has unstable angina
* Patient is in New York Heart Association functional class IV
* Patient has significant abnormality in wall motion
* Patient is affected by active endocarditis.
* Patient has a cardiac pacemaker or automatic implanted cardiac defibrillator
* Patient is affected by acute aortic dissection.
* Patient is in chronic and persistent atrial fibrillation
* Patient receives hemodialysis therapy
* Patient has a medical condition which contraindicates implantation of the SJM Epic and Epic™ Supra Porcine Bioprosthetic Heart Valve (e.g. renal failure or abnormal calcium metabolism).
* Patient has aneurysmal clips or carotid artery vascular stents
* Patient has a neurostimulator
* Patient has an implanted or external drug infusion device (e.g. insulin pump)
* Patient has a bone growth/fusion stimulator
* Patient has a cochlear, otologic, or ear implant
* Patients with severe claustrophobia in which medical sedation is contraindicated or unable to resolve anxiety sufficiently
* Patients with ocular foreign body (e.g. metal shavings)
* Patient is pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The comparison of left ventricular mass index (LVMI) at 6 months between echocardiogram (echo) and MRI in patients implanted with an Epic valve | At 6 months

CONTACTS AND LOCATIONS:
Overall Officials: G. Gerosa, Prof., Principal Investigator — Policlinico Universitario Cardiovasculare - Padua - Italy
Locations (1):
- Städtlishes Klinikum Braunschweig, Braunschweig, Germany

REFERENCES:
- [Derived] Breitenbach I, Harringer W, Tsui S, Amorim MJ, Herregods MC, Bogaert J, Goiti JJ, Gerosa G. Magnetic resonance imaging versus echocardiography to ascertain the regression of left ventricular hypertrophy after bioprosthetic aortic valve replacement: results of the REST study. J Thorac Cardiovasc Surg. 2012 Sep;144(3):640-645.e1. doi: 10.1016/j.jtcvs.2011.11.017. Epub 2011 Dec 10. PMID 22154789